CLINICAL TRIAL: NCT04648917
Title: GASC1 Inhibitor Caffeic Acid for Advanced Squamous Esophageal Cell Cancer (ESCC): a Multicenter, Phase II Trial (GiCAEC)
Brief Title: GASC1 Inhibitor Caffeic Acid for Squamous Esophageal Cell Cancer (ESCC)
Acronym: GiCAEC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Henan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GiCAEC-LY002
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Esophagus Cancer, Stage III
Keywords: esophageal cancer; caffeic acid
MeSH Terms: conditions — Esophageal Neoplasms | interventions — caffeic acid

STUDY DESIGN:
Intervention Model Description: 1:1 Randomized grouping
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): In Arm A: 40 patients will receive coffeic acid treatment: 100-200mg, tid, po, 2 weeks treated then 1 week black interval (weight >50kg, 200mg per time, weight < or =50kg, 100mg per time)
  Interventions: Drug: Caffeic acid
- Arm B (Placebo Comparator): In Arm B: 40 patients will receive the placebo tablets: 100-200mg, tid, po, 2 weeks treated then 1 week black interval.
  Interventions: Drug: Caffeic acid

INTERVENTIONS:
Drug: Caffeic acid — 40 patients will receive coffeic acid treatment: 100-200mg, tid, po, 2 weeks treated then 1 week black interval(weight >50kg, 200mg per time, weight < or =50kg, 100mg per time)

SUMMARY:
Caffeic acid can target inhibit GASC1 (gene amplified in squamous cell carcinoma 1, also known as KDM4C and JMJD2C) expression and GASC1 is confirmed to be a new oncogene in several cancers including esophageal cancer. This study aims to investigate the efficiency and safety of coffeic acid in chinese advanced esophageal squamous cell cancer (ESCC).

DETAILED DESCRIPTION:
Background: More than half of global esophageal cancer cases came from China.80 percentage patients were diagnosed with advanced disease and suffered from the poor outcome.With the development of target therapy among cancers,the overall survival and life quality of patients has been continuous improved recently.However,there had little reports focusing on target therapy in esophageal cancer . Caffeic acid as an ordinary drug is used for thrombocytopenia when patient received chemotherapy. Newly studies shown caffeic acid can target inhibit GASC1 expression, and GASC1 is confirmed to be a new oncogene in esophageal cancer.

Aim: to investigate the efficiency and safety of caffeic acid in chinese advanced esophageal squamous cell cancer.

Methods: 80 advanced ESCC patients who failed to the chemotherapy or chemoradiotherapy (1 or 2 line) will be randomized to two arms: arm A and arm B. In arm A, 40 patients will receive coffeic acid treatment: 100-200mg, tid, po, 2 weeks treated then 1 week black interval(weight >50kg, 200mg per time, weight < or =50kg, 100mg per time; in arm B, 40 patients will receive the placebo tablets. 1 years follow-up for all patients in this trial. Patients in both arms can receive any other ways of anti cancer therapy in the same time.

Primary endpoints: OS; Second endpoints: PFS

ELIGIBILITY:
Inclusion Criteria:

1. Chinese
2. esophageal squamous cell cancer
3. stage IV or recurrence disease
4. chemotherapy, or radiotherapy, or palliative care is going on

Exclusion Criteria:

1. PS (performance status): ≥ 3
2. severe hepatic and renal dysfunction
3. hypercoagulability
4. thrombocytosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | 1 year
  The percentage of 1 year overall survival (OS) after random allocation. The follow-up will be done every 3 months through phone call, investigator visiting, and medical recording review.

SECONDARY OUTCOMES:
progression-free survival (PFS) | 1 year
  The percentage of 3 months progression-free survival (PFS) after random allocation. PFS was defined as the time from randomisation to disease progression or death as assessed by the treating physicians in the study through CT scan, gastroscopy and biopsy pathology, X-ray barium meal.

CONTACTS AND LOCATIONS:
Overall Officials: Shegan Gao, Ph.D, Study Chair — The Clinical Medical College, The First Affiliated Hospital of Henan Science and Technology
Locations (3):
- China (3):
  - Anyang Tumor Hospital, Anyang, Henan
  - The Clinical Medical College, The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan

REFERENCES:
- [Result] Pedersen MT, Kooistra SM, Radzisheuskaya A, Laugesen A, Johansen JV, Hayward DG, Nilsson J, Agger K, Helin K. Continual removal of H3K9 promoter methylation by Jmjd2 demethylases is vital for ESC self-renewal and early development. EMBO J. 2016 Jul 15;35(14):1550-64. doi: 10.15252/embj.201593317. Epub 2016 Jun 6. PMID 27266524
- [Result] Movassaghian S, Xie Y, Hildebrandt C, Rosati R, Li Y, Kim NH, Conti DS, da Rocha SR, Yang ZQ, Merkel OM. Post-Transcriptional Regulation of the GASC1 Oncogene with Active Tumor-Targeted siRNA-Nanoparticles. Mol Pharm. 2016 Aug 1;13(8):2605-21. doi: 10.1021/acs.molpharmaceut.5b00948. Epub 2016 Jun 27. PMID 27223606
- [Result] Sudo G, Kagawa T, Kokubu Y, Inazawa J, Taga T. Increase in GFAP-positive astrocytes in histone demethylase GASC1/KDM4C/JMJD2C hypomorphic mutant mice. Genes Cells. 2016 Mar;21(3):218-25. doi: 10.1111/gtc.12331. Epub 2016 Jan 25. PMID 26805559
- [Result] Jia R, Yang L, Yuan X, Kong J, Liu Y, Yin W, Gao S, Zhang Y. GASC1 Promotes Stemness of Esophageal Squamous Cell Carcinoma via NOTCH1 Promoter Demethylation. J Oncol. 2019 Mar 26;2019:1621054. doi: 10.1155/2019/1621054. eCollection 2019. PMID 31031809
- [Result] Uimonen K, Merikallio H, Paakko P, Harju T, Mannermaa A, Palvimo J, Kosma VM, Soini Y. GASC1 expression in lung carcinoma is associated with smoking and prognosis of squamous cell carcinoma. Histol Histopathol. 2014 Jun;29(6):797-804. doi: 10.14670/HH-29.797. Epub 2013 Dec 27. PMID 24371038
- [Result] Sun LL, Holowatyj A, Xu XE, Wu JY, Wu ZY, Shen JH, Wang SH, Li EM, Yang ZQ, Xu LY. Histone demethylase GASC1, a potential prognostic and predictive marker in esophageal squamous cell carcinoma. Am J Cancer Res. 2013 Nov 1;3(5):509-17. eCollection 2013. PMID 24224128
- [Result] Berdel B, Nieminen K, Soini Y, Tengstrom M, Malinen M, Kosma VM, Palvimo JJ, Mannermaa A. Histone demethylase GASC1--a potential prognostic and predictive marker in invasive breast cancer. BMC Cancer. 2012 Nov 14;12:516. doi: 10.1186/1471-2407-12-516. PMID 23148692
- [Result] Jia R, Mi Y, Yuan X, Kong D, Li W, Li R, Wang B, Zhu Y, Kong J, Ma Z, Li N, Mi Q, Gao S. GASC1-Adapted Neoadjuvant Chemotherapy for Resectable Esophageal Squamous Cell Carcinoma: A Prospective Clinical Biomarker Trial. J Oncol. 2020 Jan 30;2020:1607860. doi: 10.1155/2020/1607860. eCollection 2020. PMID 32411232
- [Result] Yang ZQ, Imoto I, Fukuda Y, Pimkhaokham A, Shimada Y, Imamura M, Sugano S, Nakamura Y, Inazawa J. Identification of a novel gene, GASC1, within an amplicon at 9p23-24 frequently detected in esophageal cancer cell lines. Cancer Res. 2000 Sep 1;60(17):4735-9. PMID 10987278
- [Result] Cederblad L, Thunberg U, Engstrom M, Castro J, Rutqvist LE, Laytragoon-Lewin N. The combined effects of single-nucleotide polymorphisms, tobacco products, and ethanol on normal resting blood mononuclear cells. Nicotine Tob Res. 2013 May;15(5):890-5. doi: 10.1093/ntr/nts207. Epub 2012 Oct 4. PMID 23042982
- [Result] Yuan X, Kong J, Ma Z, Li N, Jia R, Liu Y, Zhou F, Zhan Q, Liu G, Gao S. KDM4C, a H3K9me3 Histone Demethylase, is Involved in the Maintenance of Human ESCC-Initiating Cells by Epigenetically Enhancing SOX2 Expression. Neoplasia. 2016 Oct;18(10):594-609. doi: 10.1016/j.neo.2016.08.005. Epub 2016 Sep 19. PMID 27742014